CLINICAL TRIAL: NCT00718679
Title: Evaluation of Safety, Tolerability, Immunogenicity and Efficacy of a Novel Method in Specific Immunotherapy in Cat Allergic Patients: a Placebo Controlled Trial
Acronym: IVN-CAT-001B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: ImVision GmbH, Hannover (Unknown)
Responsible Party: PD Dr. Thomas Kündig, University Hospital Zurich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVN-CAT-001B
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2010-02

CONDITIONS: Allergy to Cat Dander

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Study drug
  Interventions: Drug: IVN201
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IVN201 — Intralymphativ injection of the study drug
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
This study is placebo controlled, double blind, randomised, two arm dose escalation of a new product for specific immunotherapy in cat allergic patients

ELIGIBILITY:
Inclusion criteria:

* History and subjective symptoms of cat dander allergy including cat specific allergic rhinitis
* Age 18 to 65 years
* Positive reaction to at least one concentration of cat dander allergen in skin prick test, intradermal provocation test and nasal provocation test

Exclusion criteria:

* Chronic infectious disease
* Acute infections
* Episode of non-allergic rhinitis within the last 4 weeks
* Use of allergen known to predict anaphylactic reactions
* Treatment with any other investigational drug within 3 months before trial entry
* Vaccination within the last week
* Nasal surgery within the last 8 weeks
* Progressive fatal disease
* Drug or alcohol abuse within the last 5 years
* Cat ownership
* A history of significant cardiac insufficiency (NYHA stage III-IV)
* Coexisting severe disease, e.g. cardiovascular diseases
* Acute or history of obstructive respiratory insufficiency ( FEV1 <70%)
* Hepatic insufficiency
* Relevant anaemia (as judged by investigator)
* Blood donation within the last 30 days or intended blood donation (during the study or 30 days after participation)
* Pregnancy or breast feeding
* Sexually active woman of childbearing potential not actively practicing birth control by using a medically accepted device or therapy
* Lack of compliance or other sililar reason, that the investigator believes, precludes satisfactory participation in the study
* Systemic glucocorticoid therapy
* Allergic asthma and chronic medication with steroids at doses exceeding 200ug/day Treatment with ATII antagonists, B-blocker, ACE inhibitors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Saftety tolerability and efficacy | 2009

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Senti, MD, Principal Investigator — UniversitaetsSpital Zuerich
Locations (1):
- Center for Clinical Research University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Freiberger SN, Zehnder M, Gafvelin G, Gronlund H, Kundig TM, Johansen P. IgG4 but no IgG1 antibody production after intralymphatic immunotherapy with recombinant MAT-Feld1 in human. Allergy. 2016 Sep;71(9):1366-70. doi: 10.1111/all.12946. Epub 2016 Jun 17. PMID 27253988
- [Derived] Senti G, Crameri R, Kuster D, Johansen P, Martinez-Gomez JM, Graf N, Steiner M, Hothorn LA, Gronlund H, Tivig C, Zaleska A, Soyer O, van Hage M, Akdis CA, Akdis M, Rose H, Kundig TM. Intralymphatic immunotherapy for cat allergy induces tolerance after only 3 injections. J Allergy Clin Immunol. 2012 May;129(5):1290-6. doi: 10.1016/j.jaci.2012.02.026. Epub 2012 Mar 30. PMID 22464647